CLINICAL TRIAL: NCT01741090
Title: The Evaluation of Effectiveness and Safety for New Therapy With Bone Marrow Derived Autologous Mesenchymal Stem Cell for Hepatic Failure Caused by Alcoholic Liver Cirrhosis
Brief Title: The Effectiveness and Safety for Mesenchymal Stem Cell for Alcoholic Liver Cirrhosis
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Yonsei University (Other)
Responsible Party: Principal Investigator, Moon Young Kim, Associate Professor, Yonsei University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR109021
Record Dates: First submitted 2011-11-10; First posted 2012-12-04 (Estimated); Last update posted 2012-12-10 (Estimated); Status verified 2012-12

CONDITIONS: Alcoholic Liver Cirrhosis
Keywords: Autologous Mesenchymal stem cell; alcoholic liver cirrhosis
MeSH Terms: conditions — Liver Cirrhosis, Alcoholic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- MSC injection (Experimental): This study is designed as single interventional arm without comparative arm. MSC injection means hepatic artery catheterizations and mesenchymal stem cell injection through catheter.
  Interventions: Biological: mesenchymal stem cell injection

INTERVENTIONS:
Biological: mesenchymal stem cell injection — Hepatic artery catheterization and mesenchymal stem cell injection will be used in alcoholic liver cirrhosis. And before and 1 month after injection, change of liver cirrhosis and portal hypertension will be evaluated.

SUMMARY:
Background & Aim: Bone marrow derived mesenchymal stem cells (BM-MSCs) have capacity to differentiate into hepatocytes and anti-fibrotic effect in the experimental model. No study was done in humans with alcoholic liver cirrhosis. The researchers investigated the anti-fibrotic effect of BM-MSCs in alcoholic cirrhosis as Phase II clinical study.

Methods: Eleven alcoholic cirrhosis patients (M:F = 10:1) with Child-Pugh's class B and maintenance of alcohol abstinence at least 2 months were enrolled. At baseline, all patients received liver biopsy, hepatic venous pressure gradient (HVPG) measurement and serologic tests. BM-MSCs were isolated from each patient's BM and amplified for one month and injected two times at 4, 8week through Rt. hepatic artery. 5x106cells/mL of BM-MSCs were injected in each session. Follow up biopsy, HVPG and relative expression of tissue transforming growth factor-1 (TGF-β1), α smooth muscle actin (α-SMA) and collagen-1 by real time RT PCR were measured after 12weeks from 2nd BM-MSC injection. The primary outcome was improvement in patients' histology Aim :

The researchers aimed to evaluate safety and effectiveness of new therapy with bone marrow derived autologous mesenchymal stem cell for hepatic failure caused by alcoholic liver cirrhosis.

DETAILED DESCRIPTION:
Autologous BM-MSCs therapy in alcoholic cirrhosis induces improvement of hepatic fibrosis in histological and quantitative measurements.

ELIGIBILITY:
Inclusion Criteria:

1. Alcoholic liver cirrhosis(child Pugh class B or C, ≥ 7 scores),confirmed by clinically or biopsy.
2. Stop drinking over past 6months.
3. Patients agree with informed consent Patients must satisfy all inclusion criteria.

Exclusion Criteria:

1. Patients who did not satisfy inclusion criteria
2. Hepatocellular carcinoma
3. Pregnancy or breast feeding
4. Infective disease(HIV, HBV, HCV..)
5. Other incurable malignancy

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 12 (Estimated)
Dates: Start 2009-09; Primary Completion 2013-06 (Estimated); Study Completion 2013-08 (Estimated)

PRIMARY OUTCOMES:
The improvement of Liver Histologic grade | 6 months later
  according to Metavir and Laennec fibrosis scoring system

SECONDARY OUTCOMES:
The evaluation of hepatic dendritic cells activity by immunohistochemistry | baseline and 6 months later
Liver fibrosis quantitative analysis using Hydroxyproline contents in liver tissue | baseline and 6 months later
  Hydroxyproline is a essential component of collange fiber
Real-Time Polymerase Chain Reaction for relative mRNA expression of TGF-beta, collagen, procollagen, MMP2 or 9 | baseline and 6 months later
Hepatic venous pressure gradient(HVPG) | baseline and 6 months later
  HVPG is a gold standard to measure the portal hypertension.
Hepatic vein arrival time using microbubble contrast enhanced ultrasonography | baseline and 6 months later
  Hepatic vein arrival time is related with portal hypertension and intrahepatic inflammation, neoangiogenesis and shunts formation secondary to hepatic fibrosis.
Liver stiffness measurement with transient elastography | baseline and 6 months later
  Recently, hepatic fibrosis can be estimated non-invasively using transient elastography (Fibroscan, commercial name) and it can be additive data in estimation of therapeutic response.
Child-Pugh score | baseline and 6 months later
MELD score | baseline and 6 months later

CONTACTS AND LOCATIONS:
Overall Officials: Soon Koo Baik, M.D, Principal Investigator — Yonsei University Wonju College of Medicine Department of Internal Medicine Devision of Gastroenterology and Hepatology
Locations (1):
- Yonsei University Wonju College of Medicine Wonju Christian Hospital, Wŏnju, Gangwon-do, South Korea

REFERENCES:
- [Background] Kountouras J, Billing BH, Scheuer PJ. Prolonged bile duct obstruction: a new experimental model for cirrhosis in the rat. Br J Exp Pathol. 1984 Jun;65(3):305-11. PMID 6743531
- [Background] Batts KP, Ludwig J. Chronic hepatitis. An update on terminology and reporting. Am J Surg Pathol. 1995 Dec;19(12):1409-17. doi: 10.1097/00000478-199512000-00007. PMID 7503362
- [Background] Hong SH, Gang EJ, Jeong JA, Ahn C, Hwang SH, Yang IH, Park HK, Han H, Kim H. In vitro differentiation of human umbilical cord blood-derived mesenchymal stem cells into hepatocyte-like cells. Biochem Biophys Res Commun. 2005 May 20;330(4):1153-61. doi: 10.1016/j.bbrc.2005.03.086. PMID 15823564
- [Background] Lee KD, Kuo TK, Whang-Peng J, Chung YF, Lin CT, Chou SH, Chen JR, Chen YP, Lee OK. In vitro hepatic differentiation of human mesenchymal stem cells. Hepatology. 2004 Dec;40(6):1275-84. doi: 10.1002/hep.20469. PMID 15562440
- [Background] Kang XQ, Zang WJ, Bao LJ, Li DL, Song TS, Xu XL, Yu XJ. Fibroblast growth factor-4 and hepatocyte growth factor induce differentiation of human umbilical cord blood-derived mesenchymal stem cells into hepatocytes. World J Gastroenterol. 2005 Dec 21;11(47):7461-5. doi: 10.3748/wjg.v11.i47.7461. PMID 16437717
- [Background] Kallis YN, Alison MR, Forbes SJ. Bone marrow stem cells and liver disease. Gut. 2007 May;56(5):716-24. doi: 10.1136/gut.2006.098442. Epub 2006 Dec 4. No abstract available. PMID 17145739
- [Background] Wang JA, Luo RH, Zhang X, Xie XJ, Hu XY, He AN, Chen J, Li JH. Bone marrow mesenchymal stem cell transplantation combined with perindopril treatment attenuates infarction remodelling in a rat model of acute myocardial infarction. J Zhejiang Univ Sci B. 2006 Aug;7(8):641-7. doi: 10.1631/jzus.2006.B0641. PMID 16845718
- [Background] Kim MY, Cho MY, Baik SK, Park HJ, Jeon HK, Im CK, Won CS, Kim JW, Kim HS, Kwon SO, Eom MS, Cha SH, Kim YJ, Chang SJ, Lee SS. Histological subclassification of cirrhosis using the Laennec fibrosis scoring system correlates with clinical stage and grade of portal hypertension. J Hepatol. 2011 Nov;55(5):1004-9. doi: 10.1016/j.jhep.2011.02.012. Epub 2011 Feb 24. PMID 21354227
- [Derived] Jang YO, Kim YJ, Baik SK, Kim MY, Eom YW, Cho MY, Park HJ, Park SY, Kim BR, Kim JW, Soo Kim H, Kwon SO, Choi EH, Kim YM. Histological improvement following administration of autologous bone marrow-derived mesenchymal stem cells for alcoholic cirrhosis: a pilot study. Liver Int. 2014 Jan;34(1):33-41. doi: 10.1111/liv.12218. Epub 2013 Jun 19. PMID 23782511